CLINICAL TRIAL: NCT04627545
Title: Co-incubation of Oocytes With Sperm: Defining the Optimal Incubation Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-ABU-010-ND
Record Dates: First submitted 2020-11-03; First posted 2020-11-13 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Threshold Limit Values

STUDY DESIGN:
Intervention Model Description: Oocytes of one patient will be evenly and randomly distributed between two timings of exposure to sperm: 2h exposure versus overnight exposure (16-20h)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVF: 2h exposure (Experimental): Half of a patients' oocytes will be subjected to 2h exposure to sperm
  Interventions: Other: 2h exposure to sperm for IVF
- IVF: overnight exposure (Active Comparator): Half of a patients' oocytes will be subjected to overnight incubation with sperm (=usual practice).
  Interventions: Other: overnight exposure to sperm for IVF

INTERVENTIONS:
Other: 2h exposure to sperm for IVF — Oocytes will only be briefly (2h) exposed to progressive motile sperm for insemination
  Other Names: short exposure
  Arms: IVF: 2h exposure
Other: overnight exposure to sperm for IVF — Oocytes will be exposed for a longer duration (overnight, 16-20h) to progressive motile sperm for insemination
  Other Names: long exposure
  Arms: IVF: overnight exposure

SUMMARY:
The current pilot study aims to evaluate the fertilization rates between sibling oocytes subjected to short incubation (2h) versus overnight incubation (16-20h). As secondary objectives, the abnormal fertilization, embryo development, blastocyst biopsy and euploid rates will be analyzed.

DETAILED DESCRIPTION:
All patients for whom at least 6 cumulus oocytes complexes (COCs) are assigned to IVF, with normal sperm parameters, are eligible for the study. An electronically generated randomization list will allocate the first half of the oocytes to one arm and the other half of the oocytes to the second arm. In case an odd number of oocytes will be inseminated, one extra oocyte will be allocated to the first arm. In this prospective observational pilot study, the fertilization potential of 40 patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Sperm parameters

  * Sperm concentration before capacitation: >15 million per ml (WHO) Total motility (PR+NP %): >40 (WHO) Progressive motility (PR %):>32 (WHO)
  * Sperm concentration after capacitation: >0.6 million per ml (not WHO defined) Progressive motility (PR %):>65 (WHO)
* ≥6 COCs assigned to IVF
* BMI ≤35 kg/m2
* Female age 18 to ≤ 43 years
* All ovarian stimulation protocols
* Fresh ejaculates
* Abstinence duration 2-5 days
* Presence or absence of sperm morphology data: as we do not have a diagnostic sperm analysis for all patients, the presence or absence of >4% normal morphology (WHO) will not be taken into account, even with known low (<4%) normal morphology
* Couples requesting Preimplantation Genetic Testing for Aneuploidies
* Arab population

Exclusion Criteria:

* If the volume to be added after IVF is insufficient to perform IVF on all needed oocytes
* Presence of >1 million per ml round cells in the ejaculate
* If a couple's previous cycle was included in the study
* Previous history of fertilization failure or <50% fertilisation
* Globozoospermia
* PCO according to the Rotterdam criteria
* Progesterone >1.5 ng/ml on the day of trigger

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female patients seeking fertility treatment
Enrollment: 55 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Normal fertilization rate | 2 days
  presence of two pronuclei per inseminated oocyte

SECONDARY OUTCOMES:
Number of COCs assigned to each group | 2 days
  number of oocytes, per patient, assigned to each exposure group
Maturation rate | 2 days
  number of mature oocytes obtained in each arm
Fertilization | 3 days
  Number of abnormally fertilized oocytes and failed fertilization
Total fertilization failure | 3 days
  Number of cycles with complete fertilization failure (in one arm or in both arms)
Embryo quality on day 3 | 5 days
  defined by the Istanbul consensus (Alpha Scientists, 2011) The number of blastomeres and their division pattern, fragmentation, presence of compaction, vacuoles, granulation and nuclei will divide the embryos into 3 categories: good, fair or poor
Embryo quality on day 5 | 8 days
  defined by a modified model of Gardner and Schoolcraft,1999
blastulation rate I | 8 days
  number of embryos reaching at least the BL1 stage/ number of oocytes assigned to that group: defined by a 1 (yes, the embryo is blastulating) or 0 (no, the embryo is not blastulating)
blastulation rate II | 8 days
  number of embryos reaching at least the BL1 stage/ number of mature oocytes in that group: defined by a 1 (yes, the embryo is blastulating) or 0 (no, the embryo is not blastulating)
Utilization rate | 8 days
  number of embryos that can be used for the patient (=number of embryos that can be biopsied)/number of oocytes assigned to the group
Day of trophectoderm biopsy | 8 days
  Day at which the blastocyst reaches sufficient expansion to perform biopsy of trophectoderm cells
Euploid rate | 8 days
  Number of genetically normal embryos per total number of blastocysts biopsied, stratified per day of biopsy
Morphokinetic parameters | 10 days
  As embryos will be monitored in a time lapse imaging system, morphokinetic parameters will be compared between both exposure arms: o t2: the timing to two cells
  * t3: the timing to three cells
  * t4: the timing to four cells
  * t5: the timing to five cells
  * t8: the timing to eight cells
  * SC: starting to compact
  * M: the timing to morula
  * SB: starting to blastulate
  * B: reaching a BL3 according to Gardner and Schoolcraft, 1999
  * F: reaching a BL4 according to Gardner and Schoolcraft, 1999
  * cc2: t3-t2
  * s2: t4-t3
Pregnancy outcome | 60 days
  dichotomous variable defined by the presence of βhCG test of > 15IU 12-15 days after embryo transfer
Biochemical pregnancy | 70 days
  dichotomous variable defined as a pregnancy in which the hCG levels start do decrease after 1 week
Implantation rate | 80 days
  defined by the number of gestational sacs/number of embryos transferred
  • Clinical pregnancy (yes or no) defined by the ultrasonographic visualization of one or more gestational sacs, including ectopic pregnancies
Clinical pregnancy Fetal Heart beat positive | 80 days
  dichotomous variable defined by the ultrasonographic visualization of one or more gestational sacs, with fetal heart beat at 7 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Neelke De Munck, PhD, Principal Investigator — ART Fertility Clinics
Locations (1):
- ART Fertility Clinics, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
The principal investigator will gather all data for the study and prepare the database for the statistician, who will be blinded for patient information.